CLINICAL TRIAL: NCT05584150
Title: Assessment of the Benefit of a Deep Cleansing Gel Containing Salicylic Acid 2%, Zinc Gluconate 0.2% and Lipohydroxy Acids 0.05% in Patients With Mild to Moderate Truncal Acne: Results From an Exploratory Study
Brief Title: The Benefit of a Deep Cleansing Gel in the Management of Mild to Moderate Truncal Acne
Status: Completed | Type: Observational
Sponsor: Cosmetique Active International (Industry)
Responsible Party: Sponsor
Other Study IDs: 1819CBCL747
Record Dates: First submitted 2022-09-25; First posted 2022-10-18 (Actual); Last update posted 2022-10-18 (Actual); Status verified 2022-09

CONDITIONS: Acne
Keywords: truncal acne
MeSH Terms: conditions — Acne Vulgaris

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Deep Cleansing Gel — daily use

SUMMARY:
Acne vulgaris is a chronic inflammatory disease, mainly of the face, but also of the trunk. Acne may be caused by internal and external factors. Only a very small amount of data exists concerning truncal acne. The condition affects about 9% of the population worldwide, with 50% of subjects with facial acne also presenting with truncal acne. Until recently, clinicians frequently followed the same therapeutic approach as for facial acne, with treatment adherence remaining an issue.

This study assessed assessed the benefit of a cleansing gel containing salicylic acid 2%, zinc gluconate 0.2% and Lipo hydroxy acids (LHA) 0.05%, used daily for 84 days in mild to moderate truncal acne.

DETAILED DESCRIPTION:
For this single center, open label, non-randomized exploratory study, 51 subjects with mild to moderate truncal acne were recruited. The study received ethics committee approval. All subjects provided written informed consent. The investigator evaluated the number of inflammatory, non-inflammatory and total lesions at Baseline, Day 42 and 84. Skin barrier function was appraised via the assessment of transepidermal water loss (TEWL) using a Tewameter® (Courage + Khazaka Electronic GmbH, Germany). Safety was assessed by considering the evaluation of clinical signs and reporting of symptoms, and local adverse reactions. Subjects were asked to gently massage the wet skin of the trunk with the product in the morning and evening for at least 30 seconds, and then thoroughly rinse with tempered water and pat dry.

ELIGIBILITY:
Inclusion Criteria:

* above 18 years
* truncal acne

Exclusion Criteria:

- None

Ages: 18 Years to 99 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: adult female or males with subjects with truncal acne
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2020-11-30 (Actual)

PRIMARY OUTCOMES:
Investigator global assessment | baseline
  Scale 0=absent to 5=very serious
Investigator global assessment | Day 42
  Scale 0=absent to 5=very serious
Investigator global assessment | Day 84
  Scale 0=absent to 5=very serious

SECONDARY OUTCOMES:
inflammatory lesion count | baseline
  count and percentage reduction
inflammatory lesion count | Day 42
  count and percentage reduction
inflammatory lesion count | Day 84
  count and percentage reduction
non-inflammatory lesion count | baseline
  count and percentage reduction
non-inflammatory lesion count | Day 42
  count and percentage reduction
non-inflammatory lesion count | Day 84
  count and percentage reduction
total lesion count | baseline
  count and percentage reduction
total lesion count | Day 42
  count and percentage reduction
total lesion count | Day 84
  count and percentage reduction
acne severity | baseline
  scale 0=absent to 5=very severe
acne severity | Day 42
  scale 0=absent to 5=very severe
acne severity | Day 84
  scale 0=absent to 5=very severe
transepidermal water loss | baseline
  tewameter assessment
transepidermal water loss | Day 42
  tewameter assessment
transepidermal water loss | Day 84
  tewameter assessment
clinical safety | baseline
  assessment of clinical signs symptoms and adverse events
clinical safety | Day 42
  assessment of clinical signs symptoms and adverse events
clinical safety | Day 84
  assessment of clinical signs symptoms and adverse events
subject efficacy perception | Day 42
  scale 0=none to 5= very good
subject efficacy perception | Day 84
  scale 0=none to 5= very good
subject product perception | Day 84
  sacle 0=bad to 5 very good

CONTACTS AND LOCATIONS:
Overall Officials: Delphine Kerob, MD, Study Director — La Roche-Posay Laboratoire Dermatologique
Locations (1):
- CIDP, Rio de Janeiro, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Towersey L, Correia P, Fajgenbaum Feiges M, Euzebio Goncalves Junior J, Sant'Anna B, Kerob D, Le Floc'h C. Assessment of the Benefit of a Deep Cleansing Gel Containing Salicylic Acid 2%, Zinc Gluconate 0.2% and Lipohydroxy Acids 0.05% in Patients with Mild to Moderate Truncal Acne: Results from an Exploratory Study. Clin Cosmet Investig Dermatol. 2023 Jan 18;16:119-123. doi: 10.2147/CCID.S394123. eCollection 2023. PMID 36698447